CLINICAL TRIAL: NCT03099785
Title: A Phase II, Multicentre, Randomised, Double-blind, Placebo Controlled, Proof of Concept Study of Efficacy and Safety of Rifamycin SV-MMX® 600 mg Tablets Administered Three or Two Times Daily to Patients With Diarrhoea-predominant Irritable Bowel Syndrome (IBS-D)
Brief Title: Rifamycin SV-MMX® 600 mg Tablets Administered Three or Two Times Daily to Patients With IBS-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cosmo Technologies Ltd (Industry)
Responsible Party: Sponsor
Organization: Cosmo Pharmaceuticals NV (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CB-01-11/28
Record Dates: First submitted 2017-03-14; First posted 2017-04-04 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Diarrhea-predominant Irritable Bowel Syndrome
MeSH Terms: interventions — rifamycin SV

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment group 1: dose regimen 1 (Active Comparator): Rifamycin SV-MMX® 600 mg modified release tablets, three times daily (t.i.d.)
  Interventions: Drug: Rifamycin SV 600mg t.i.d.
- Treatment group 2: dose regimen 2 (Active Comparator): Rifamycin SV-MMX® 600 mg modified release tablets, two times daily (b.i.d.) + matching placebo daily (q.d.)
  Interventions: Drug: Rifamycin SV b.i.d. + Placebo
- Treatment group 3: matching placebo (Placebo Comparator): Rifamycin SV-MMX® matching placebo tablets, t.i.d.
  Interventions: Drug: Placebo t.i.d.

INTERVENTIONS:
Drug: Rifamycin SV 600mg t.i.d. — Morning: one 600 mg tablet Afternoon: one 600 mg tablet Evening: one 600 mg tablet
  Arms: Treatment group 1: dose regimen 1
Drug: Rifamycin SV b.i.d. + Placebo — Morning. one 600 mg tablet Afternoon: one matching placebo tablet Evening: one 600 mg tablet
  Arms: Treatment group 2: dose regimen 2
Drug: Placebo t.i.d. — Morning. one matching placebo tablet Afternoon: one matching placebo tablet Evening: one matching placebo tablet
  Arms: Treatment group 3: matching placebo

SUMMARY:
The objective of this study is to evaluate the safety and efficacy Rifamycin SV-MMX® 600 mg tablets for patients with diarrhoea-predominant irritable bowel syndrome when administered two to three times daily.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent: signed written informed consent before inclusion in the study
2. Sex and Age: males/females, ≥18 year old
3. IBS Diagnosis: confirmed IBS-D diagnosis per Rome IV criteria
4. Symptoms: active symptoms of IBS at baseline (day 1) as measured by average daily scores for at least 7 days before baseline:

   1. abdominal pain score ≥3 using an 11-point numeric rating scale and
   2. bloating score: 2-4 inclusive and
   3. stool consistency: score 6 or 7 (measured by the Bristol stool form scale) for at least 2 days from day -7 to day -1

      and by a negative response to the global IBS symptom assessment question and to the IBS-related bloating assessment question both given weekly during the screening phase up to day 1 before randomisation:
   4. "In the past 7 days, have you had adequate relief of your IBS symptoms?" [No] and
   5. "In the past 7 days, have you had adequate relief of your IBS symptom of bloating?"[No]
5. Colonoscopy: performed within 5 years; if patient's age >50, colonoscopy performed within 2 years
6. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the study
7. Literacy: sufficiently literate to comply with the study requirement of using electronic diaries and filling in electronic forms
8. Contraception and fertility: females of childbearing potential and fertile males must be using at least one reliable method of contraception.

Reliable methods of contraception for women include:

1. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit
2. A non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit

   Reliable methods of contraception for men and male partners of female patients include:
3. Male condoms with spermicide

   Reliable methods of contraception for both women and men include:
4. A sterile sexual partner or sexual abstinence Women of non-childbearing potential or in post-menopausal status for at least 1 year and sterile or surgically sterilised men will be admitted.

For women of childbearing potential, serum pregnancy test result must be negative at screening

Exclusion Criteria:

1. IBS: symptoms of constipation at baseline:

   1. less than 3 bowel movements a week and
   2. stool consistency score ≤2 for ≥2 days in a week
2. Screening phase: failure to record the daily symptom assessments in the diary cards for at least 7 days before baseline
3. Gastroenteric: underlying gastrointestinal diseases including ulcerative colitis, Crohn's disease, pancreatitis, any active infectious, haemorrhagic or inflammatory disorder not related to IBS-D, gastrointestinal motility disorders such as ileus, gastroparesis or pseudoobstruction, gastroduodenal ulcer, gastrointestinal malignancy or potentially fatal diseases if not full in remission (5 years from diagnosis and without maintenance treatment), amyloidosis and cholelithiasis if cholecystectomy not performed
4. Intolerance: ascertained underlying lactose intolerance with response to diet or any other malabsorption syndrome with the exclusion of asymptomatic lactose malabsorption
5. Coeliac disease: ascertained or presumptive underlying coeliac disease
6. Bile: ascertained or presumptive bile acid malabsorption or bile acid induced diarrhoea
7. Diabetes: underlying diabetes type I or II
8. Thyroid: abnormal thyroid function not controlled by thyroid medications
9. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study
10. Renal function: ascertained or presumptive clinically significant renal insufficiency or creatinine above twice the upper limit of normal (ULN) of the performing laboratory reference range
11. Liver function: chronic liver disease or clinically significant liver enzyme abnormality as evidenced by elevated AST, ALT or total bilirubin >1.5 times ULN
12. AIDS/HIV: ascertained or presumptive acquired immunodeficiency (AIDS) or known infection with human immunodeficiency virus (HIV)
13. Diseases: significant history of medical or surgical conditions excluding hysterectomy, caesarean section, appendectomy, cholecystectomy, benign polypectomy and inguinal hernia and including renal, hepatic, cardiovascular, haematological, endocrine, immune, psychiatric or neurological diseases that in the investigator's opinion may interfere with the aim of the study; malignant diseases not in remission for at least 5 years
14. Medications: alosetron, eluxadoline, ondansetron, tegaserod, lubiprostone, warfarin, antipsychotic, antispasmodic, prokinetic, antidiarrhoeal, laxative, probiotic, narcotic or antibiotic agents within 14 days before the screening visit; antidepressant agents of the selective serotonin-reuptake inhibitor and tricyclic classes unless taken at a stable dose for at least 6 weeks before the screening visit
15. Investigational drugs: participation in the evaluation of any investigational product within 30 days before this study
16. Drug and alcohol: known history of drug or alcohol [>1 drink/day for females and >2 drinks/day for males, defined according to the USDA Dietary Guidelines 2015] abuse
17. Pregnancy (females only): pregnant or lactating women or wishing to become pregnant in the 3 months following this visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with relief from abdominal pain and improved stool consistency. | 88 days
  Proportion of weekly responders defined as subjects who weekly have relief of the composite of abdominal pain and stool consistency, on the basis of their daily assessments. Relief of abdominal pain is defined as a decrease in the weekly average of abdominal pain score of at least 30% compared with baseline and relief of stool consistency is defined as a 50% or greater reduction in the number of days per week with at least one stool that has a consistency of Type 6 or 7 compared with baseline.
  All participants will complete daily assessments of abdominal pain and stool consistency:
  * Abdominal Pain: Scored between 0 (no pain) and 10 (as bad as it could be)
  * Stool Consistency: Bristol Stool Scale (Scored 1-7)

SECONDARY OUTCOMES:
Proportion of subjects with relief of global IBS symptoms during weeks 3-12 [Efficacy] | 10 weeks
  Proportion of subjects with adequate relief of global IBS symptoms for at least 2 (consecutive or not) of the 10 weeks during the follow-up period (i.e., weeks 3 through 12). Adequate relief of global IBS symptoms is defined as a response of "yes" to the following question, which will be asked weekly (every 7 days): "In regard to all your symptoms of IBS, as compared to the way you felt before you started study medication, have you, in the past 7 days, had adequate relief of your IBS symptoms? [Yes/No]"
Proportion of subjects with monthly relief of global IBS symptoms [Efficacy] | 88 days
  Proportion of subjects with adequate relief of global IBS symptoms during at least 2 weeks (consecutive or not) per month ("monthly response") during month 1, during month 1 through 2 and during month 1 through 3 will be assessed to identify the onset and duration of the therapeutic effect.
Proportion of subjects with relief of IBS-related bloating during weeks 3-12 [Efficacy] | 10 weeks
  Proportion of subjects with adequate relief of IBS-related bloating for at least 2 (consecutive or not) of the 10 weeks during the follow-up period (i.e., weeks 3 through 12). Adequate relief of bloating is defined as a response of "yes" to the following question, which will be asked weekly (every 7 days): "In regard to your symptom of bloating, as compared to the way you felt before you started study medication, have you, in the past 7 days, had adequate relief of your IBS symptom of bloating? [Yes/No]."
Proportion of subjects with monthly relief of IBS-related bloating [Efficacy] | 88 days
  Proportion of subjects with adequate relief of bloating during at least 2 weeks (consecutive or not) per month ("monthly response") during month 1, during month 1 through 2 and during month 1 through 3 will be assessed to identify the onset and duration of the therapeutic effect.
Proportion of subjects with weekly relief of IBS symptoms, bloating and abdominal pain [Efficacy] | 88 days
  Proportion of subjects with relief (weekly responders) determined from the subjects' daily assessments of IBS symptoms, bloating, and abdominal pain; relief of IBS symptoms and bloating is defined as a score of either 0 (not at all) or 1 (hardly) for at least 50% of the days in a given week or a score of 0 (not at all), 1 (hardly), or 2 (somewhat) for 100% of the days in a given week for at least 2 (consecutive or not) of the 4 weeks during a given month. Relief of abdominal pain is defined as a decrease by ≥30% from baseline in weekly mean rating of IBS-related abdominal pain.
  All participants will complete daily assessments of IBS symptoms, bloating and abdominal pain:
  * IBS Symptoms: Scored between 0 (Not bothersome at all) and 6 (a very great deal bothersome)
  * Bloating: Scored between 0 (not at all bothersome) and 6 (a very great deal bothersome)
  * Abdominal Pain: Scored between 0 (no pain) and 10 (as bad as it could be)
Number of weeks of IBS-symptom relief during follow-up [Efficacy] | 10 weeks
  Number of weeks (consecutive or not) subjects achieve adequate relief of IBS symptoms during the follow up period.
Number of weeks of bloating relief during follow-up [Efficacy] | 10 weeks
  Number of weeks (consecutive or not) subjects achieve adequate relief of bloating during the follow up period.
Change in IBS-symptoms, bloating and abdominal pain from baseline to 12 weeks - captured by a daily diary [Efficacy] | 12 weeks
  Change from baseline to week 12 in daily IBS symptoms, bloating and abdominal pain. This information will be captured in a daily diary by the participants.
  All participants will complete daily assessments of IBS symptoms, bloating and abdominal pain:
  * IBS Symptoms: Scored between 0 (Not bothersome at all) and 6 (a very great deal bothersome)
  * Bloating: Scored between 0 (not at all bothersome) and 6 (a very great deal bothersome)
Proportion of monthly responders for IBS-symptoms, bloating and abdominal pain [Efficacy] | 3 months
  Proportion of monthly responders during month 1, during month 1 through 2 and during month 1 through 3 determined from the subjects' daily assessments of IBS symptoms, bloating, and abdominal pain; relief of IBS symptoms and bloating is defined as a score of either 0 (not at all) or 1 (hardly) for at least 50% of the days in a given month or a score of 0 (not at all), 1 (hardly), or 2 (somewhat) for 100% of the days in a given month. Relief of abdominal pain is defined as a decrease by ≥30% from baseline in weekly mean rating of IBS-related abdominal pain. Relief of stool consistency is defined as a 50% or greater reduction in the number of days per month with at least one stool that has a consistency of Type 6 or 7 compared with baseline.
  Daily Assessments:
  * IBS Symptoms: Scored between 0 (Not bothersome at all) and 6 (a very great deal bothersome)
  * Bloating: Scored between 0 (not at all bothersome) and 6 (a very great deal bothersome)
Change from baseline to each week during follow up for IBS-symptoms bloating, abdominal pain, stool consistency, urgency - captured by a daily diary [Efficacy] | 12 weeks
  Change from baseline to each week during the 12 week follow up for daily IBS symptoms, bloating, abdominal pain, stool consistency and sense of urgency, asked as "Have you felt or experienced a sense of urgency today? [Yes/No]" and calculated as 100* (number of days with urgency/number of days with data), and daily number of stools. This information will be captured in a daily diary by the participants.
  All participants will complete daily assessments of IBS symptoms, bloating and abdominal pain:
  * IBS Symptoms: Scored between 0 (Not bothersome at all) and 6 (a very great deal bothersome)
  * Bloating: Scored between 0 (not at all bothersome) and 6 (a very great deal bothersome)
  * Stool Consistency: Bristol Stool Scale (Scored 1-7)
  * Urgency: Answered Yes or No
Change from baseline at weeks 4, 8 and 12 in quality of life assessment [Efficacy] | 12 weeks
  Change from baseline at weeks 4, 8 and 12 in quality of life inquired as IBS-QoL

OTHER OUTCOMES:
Treatment Emergent Adverse Events [Safety] | 12 weeks
  Monitoring of treatment emergent adverse events.
Change from Baseline in Physical Exam [Safety] | 12 weeks
  Changes from baseline in physical examination.
Change from Baseline in Vital Signs [Safety] | 12 weeks
  Changes from baseline in vital signs.
Change from Baseline in Lab Tests [Safety] | 12 weeks
  Changes from baseline in clinical laboratory tests.
Change from Baseline in ECG [Safety] | 12 weeks
  Changes from baseline in ECG.

CONTACTS AND LOCATIONS:
Locations (29):
- Belgium (5):
  - University Hospital Gasthuisberg, Department of Gastroenterology, Leuven, Herestraat 49
  - St Lukas Ziekenhuis,, Bruges, Lucaslaan 29
  - Clinique universitaires Saint-Luc Gastroenterologie Route 606 Avenue Hippocrate, 10, Brussels
  - Maria Middelares, Digestief Centrum, Buitenring St-Denijs 30, Ghent
  - University Hospital Gent, Depintelaan 185, Ghent
- Germany (11):
  - Emovis GmbH Wilmersdorfer Straße 79, Berlin
  - Unterfrintroper Hausarztzentrum Lehrpraxis der Universität Essen, Essen
  - Internistenzentrum Bahnhofstrasse 30, Gauting
  - Clinical Research Hamburg GmbH, Rahlstedter Bahnhofstraße 33, Hamburg
  - Gastroenterologie, Interventionelle Endoskopie, Diabetologie und Akutgeriatrie, KRH-Zentrumsgeschaftsfuhrer innere Medizin, KRK Klinikum Siloah-Oststadt-Heidehaus Stadionbrucke 4, Hanover
  - Gemeinschaftspraxis Dr. Klein & J. Minnich, Künzing
  - AmBeNet GmbH, Wilhelm-Leuschner-Platz I2,, Leipzig
  - Universitatsklinikum Magdeburg A.O.R. Klinik fur Gastroenterologie, Hepatologie und Infektiologie, Leipziger Str.44, Magdeburg
  - Ärztehaus Reinfeld Praxisgemeinschaft für Allgemeinmedizin Klosterstraße 7, Reinfeld
  - Innomed Dr. med. Naudts Ludwig-Erhard-Platz 11, Rodgau
  - Internistische Praxisgemeinschaft, Bereich Gastroenterologie Hauptstraße. 51, Weyhe
- Italy (8):
  - S.O.C Gastroenterologia Oncologica, Aviano, PN
  - Azienda Ospedaliera G. Brotzu, U.O. di Gastroenterelogia, Via Peretti, Cagliari
  - Istituto Clinico Humanitas, Centro Malattie Infiammatorie Croniche Intestinali, Milan
  - Fonazione IRCCS Ospedale Maggiore, Milan
  - Fondazione IRCCS Policlinico S. Matteo, Dip Area Medica: Medicina Generale 1, Viale Camillo Golgi, 19, Pavia
  - Polo Scienze Gastroenterologiche ed, Roma
  - Universita Campus Bio Medico, U.O.C di Gastroenterologia ed Endoscopia Digestiva, Roma
  - IRCCS Policlinico San Donato, Medicina Generale III- Gastroenterologia, San Donato Milanese
- Spain (5):
  - Hospital Universitari Germans Trias i Pijol (Can Ruti). Servicio de Aparto Digestivo Carretera de Canyet, s/n, Badalona, Barcelona
  - Hospital Universitario La Paz, Servicio de Aparato Digestivo Po de la Castellana 261, Castellana, Madrid
  - Hospital Universitario Ramon Y Cajal, Servicio de Gastroenterologia y Hepatologia Ctra. de colmenar Viejo, Km 9,100, Colmenar Viejo, Madrid
  - Hospital Universitari vall d'Hebron, Servicio de Aparato Digestivo, Passeig Vall d'Hebron, 119-129, Barcelona
  - Hospital Universitario Clinico San Carlos, Servicio de Aparato Digestivo, Calle del Prof Martin Lagos, s/n,, Madrid

IPD SHARING:
Plan to Share IPD: No
None. IPD not to be shared.